CLINICAL TRIAL: NCT02273063
Title: 5Hz Repetitive Transcranial Magnetic Stimulation for Posttraumatic Stress Disorder Comorbid With Major Depressive Disorder
Brief Title: rTMS for PTSD Comorbid With Major Depressive Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Butler Hospital (Other)
Collaborators: Providence VA Medical Center (U.S. Federal Agency); Neuronetics (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1404-005
Record Dates: First submitted 2014-10-15; First posted 2014-10-23 (Estimated); Results first posted 2018-10-04 (Actual); Last update posted 2018-10-04 (Actual); Status verified 2018-10

CONDITIONS: Posttraumatic Stress Disorder; Major Depressive Disorder; Transcranial Magnetic Stimulation, Repetitive
Keywords: PTSD; MDD; TMS; 5Hz
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depressive Disorder, Major | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Transcranial Magnetic Stimulation (Experimental): Stimulation at pulse frequency of 5Hz delivered over L DLPFC. Intensity: 120% of Motor Threshold, 5 Sec Train, 14 Sec Inter-Train Interval, Frequency: 5Hz, Total Pulses: 3000/session. Sessions delivered once/day on weekdays for up to 40 sessions.
  Interventions: Device: Transcranial Magnetic Stimulation (TMS)

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation (TMS) — Up to 40 sessions of TMS delivered with the first 35 sessions delivered over 7 weeks, and final 5 treatments delivered in taper schedule over 3 weeks. Treatment is adjunct to ongoing stable pharmacotherapy.
  Other Names: Neuronetics' NeuroStar TMS Therapy System

SUMMARY:
The purpose of this study is to see how well a treatment called "Repetitive Transcranial Magnetic Stimulation" works for patients who struggle with symptoms of both posttraumatic stress disorder and major depressive disorder.

DETAILED DESCRIPTION:
This study aims to evaluate the safety and efficacy of repetitive transcranial magnetic stimulation (rTMS) for adults with comorbid posttraumatic stress disorder (PTSD) and major depressive disorder (MDD). Although standard rTMS uses stimulations delivered to the left prefrontal cortex at 10 pulses per second, prior work has shown that other stimulation frequencies may work for both PTSD and MDD. In this study, we examine the efficacy of left-sided 5Hz in patients with PTSD and MDD, hypothesizing that this lower frequency will improve PTSD and MDD symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. To ensure subjects can safely receive rTMS, eligible subjects must meet all established screening criteria for safety during MRI (magnetic resonance imaging), since MRI involves magnetic fields at similar intensity to those emitted from the rTMS treatment coil. These are conservative measures require a patient not having the following (unless MRI-safe): Cardiac pacemaker, implanted device (deep brain stimulation) or metal in the brain, cervical spinal cord, or upper thoracic spinal cord;
2. Outpatients 18-70 years of age (inclusive)
3. Meet DSM-IV criteria for MDD (recurrent or single episode chronic) and PTSD (acute or chronic) at the time of the screening and baseline visits;
4. Have a baseline score of "Moderately Ill" or worse on both the CGI-S and the PGI-S.
5. Have failed at least one antidepressant medication trial as part of definitive and adequate treatment in the current episode, OR have demonstrated intolerance to at least one antidepressant medication as part of attempted treatment in the current episode of illness (i.e., meet FDA labeling requirements for administration of rTMS for depression);
6. Be on a stable psychotropic regimen for at least six weeks (42 days) prior to screening, or no psychotropic medication at all, and be willing to maintain the current regimen and dosing for the duration of the study (unless medical necessary to make changes with notification of research staff);
7. If female and of child bearing potential, agree to use an acceptable method of birth control for the duration of the study treatment period
8. Be willing and able to comply with all study related procedures and visits,
9. Be capable of independently reading and understanding patient information materials and giving written informed consent.

Exclusion Criteria:

1. Are pregnant or lactating or planning to become pregnant within the next three months.
2. Have a lifetime history of loss of consciousness due to head injury for greater than 10 minutes, or any lifetime history of loss of consciousness due to a head injury with documented evidence of brain injury (including brain atrophy).
3. Current (or past if appropriate) significant neurological disorder, or lifetime history of a) seizure disorder b) primary or secondary CNS tumors c) stroke or d) cerebral aneurysm;
4. Current Axis 1 primary psychotic disorder, or bipolar I disorder, current alcohol and/or substance dependence or abuse within the past 1 month;
5. Past treatment with TMS therapy
6. Have active suicidal intent or plan as detected on screening assessments, or in the Investigator's opinion, is likely to attempt suicide within the next six months.
7. Demonstrate the presence of any other condition or circumstance that, in the opinion of the investigator, has the potential to prevent study completion and/or to have a confounding effect on outcome assessments.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-10; Primary Completion 2016-04-22 (Actual); Study Completion 2016-04-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linda L Carpenter, M.D., Principal Investigator — Butler Hospital
Locations (2):
- United States (2):
  - Butler Hospital, Providence, Rhode Island
  - Providence VA Medical Center, Providence, Rhode Island

REFERENCES:
- [Derived] Carpenter LL, Conelea C, Tyrka AR, Welch ES, Greenberg BD, Price LH, Niedzwiecki M, Yip AG, Barnes J, Philip NS. 5 Hz Repetitive transcranial magnetic stimulation for posttraumatic stress disorder comorbid with major depressive disorder. J Affect Disord. 2018 Aug 1;235:414-420. doi: 10.1016/j.jad.2018.04.009. Epub 2018 Apr 5. PMID 29677606
- [Derived] Philip NS, Barredo J, van 't Wout-Frank M, Tyrka AR, Price LH, Carpenter LL. Network Mechanisms of Clinical Response to Transcranial Magnetic Stimulation in Posttraumatic Stress Disorder and Major Depressive Disorder. Biol Psychiatry. 2018 Feb 1;83(3):263-272. doi: 10.1016/j.biopsych.2017.07.021. Epub 2017 Aug 8. PMID 28886760
- See also: Online ahead of print article with all methods and results — https://doi.org/10.1016/j.jad.2018.04.009

RESULTS

PARTICIPANT FLOW:
Groups:
- TMS Prescription: 5Hz delivered over L DLPFC. Intensity: 120% of Motor Threshold, 5 Sec Train, 14 Sec Inter-Train Interval, Frequency: 5Hz, Total Pulses: 3000
  Transcranial Magnetic Stimulation: Stimulating DLPFC at 5 Hz for up to 40 treatment sessions overall. 35 sessions delivered over 7 weeks, and final 5 treatments delivered in taper over 3 weeks. There will be a post treatment assessment 72 hours after final treatment, and then again 1 month after the final treatment.
Period: Overall Study
Arm/Group | TMS Prescription
Started | 40
Completed | 35
Not Completed | 5

BASELINE CHARACTERISTICS:
Population: Comorbid PTSD & MDD
Arm/Group | TMS Prescription
Number analyzed (Participants) | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.6 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 21
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 33
  Black | 1
  Multiracial | 1
Region of Enrollment [Number; unit: participants]
  United States | 35

OUTCOME MEASURES:

1. Primary Outcome: Total Score on PTSD Checklist for DSM-5 (PCL-5)
Description: This self-report scale is called: "PTSD Checklist for DSM-5" (abbreviated PCL-5) (see https://www.ptsd.va.gov/professional/assessment/adult-sr/ptsd-checklist.asp). Total PCL-5 score ranges from 0 to 80. Analysis of treatment effect on symptom severity will be evaluated by change in PCL-5 total score from baseline (pre-TMS) to endpoint (post-TMS)(or LOCF); Paired t-test compares the mean total PCL-score for the group at the two time points. A higher total score on the PCL-5 scale corresponds with more severe PTSD symptoms than a lower total score. A greater change from baseline to endpoint would correspond with better treatment outcome.
Time Frame: Baseline to final TMS session (up to 40 sessions over up to 8 weeks)
Population: intent-to-treat population
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Transcranial Magnetic Stimulation (TMS): TMS 5Hz delivered over L DLPFC. Intensity: 120% of Motor Threshold, 5 Sec Train, 14 Sec Inter-Train Interval, Frequency: 5Hz, Total Pulses: 3000
  Transcranial Magnetic Stimulation: Stimulating DLPFC at 5 Hz for up to 40 treatment sessions overall. 35 sessions delivered over 7 weeks, and final 5 treatments delivered in taper over 3 weeks. There will be a post treatment assessment 72 hours after final treatment, and then again 1 month after the final treatment.
Arm/Group | Transcranial Magnetic Stimulation (TMS)
Number analyzed (Participants) | 35
units on a scale
  BASELINE | 52.2 (13.1)
  ENDPOINT | 34.0 (21.6)

2. Primary Outcome: Total Score on Inventory of Depressive Symptomatology, Self-Report (IDS-SR) Scale
Description: This self-report scale is called "Inventory of Depressive Symptomatology, Self-Report" (Abbreviated IDS-SR). IDS-SR Total Scores Range from 0 to 84, with a higher score reflecting greater depressive symptom severity. Paired t-test compares the change in mean total IDS-SR score from baseline (pre-TMS) to endpoint (last TMS session) or LOCF. A greater change reflects a better outcome than lesser change.
Time Frame: Baseline to final TMS session (up to 40 sessions over up to 8 weeks)
Population: intent-to-treat population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TMS Prescription
Number analyzed (Participants) | 35
units on a scale
  BASELINE | 47.8 (11.9)
  ENDPOINT | 30.9 (18.9)

ADVERSE EVENTS:
Time Frame: baseline to endpoint (week 10 or LOCF).
Description: Adverse event data collected through (1) Response of participants to queries by study clinicians during treatment sessions and during study-specific assessment visits (2) spontaneous reports initiated by participants.
Arm/Group | TMS Prescription
Serious Adverse Events (participants affected / at risk) | 4/35
Other Adverse Events (participants affected / at risk) | 15/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TMS Prescription (N=35)
Psychiatric Hospitalization (Psychiatric disorders) | 4 (4)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TMS Prescription (N=35)
migraine (Nervous system disorders) | 1 (1)
Activation/insomnia/irritability (Psychiatric disorders) | 14 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No